CLINICAL TRIAL: NCT06185764
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled Single- and Multiple-dose Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VX-670 in Adult Subjects With Myotonic Dystrophy Type 1
Brief Title: A Phase 1/2 Study of VX-670 in Adult Participants With Myotonic Dystrophy 1 (DM1)
Acronym: Galileo
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX23-670-001; 2023-506028-10-00 (Other: EUCT Number)
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
Keywords: DM1; DM2; Myotonic Dystrophy 1; Myotonic Dystrophy 2; Myotonic Dystrophy Type 1 (DM1); Myotonic Dystrophy; DM; Myotonia; Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; Vertex; Entrada; VX-670; VX670; PMO; ASO; Myotonic Muscular Dystrophy; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Muscular Dystrophies
MeSH Terms: conditions — Myotonic Dystrophy; Myotonia; Myotonic Disorders; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Single Ascending Dose (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-670.
  Interventions: Drug: VX-670
- Part A: Placebo (Placebo Comparator): Participants will be randomized to receive single dose of placebo matched to VX-670.
  Interventions: Drug: Placebo
- Part B: Single and Multiple Ascending Dose (Experimental): Participants will be randomized to receive single and multiple doses of different dose levels of VX-670. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-670
- Part B: Placebo (Placebo Comparator): Participants will be randomized to receive single or multiple doses of placebo matched to VX-670.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-670 — Solution for intravenous administration.
  Arms: Part A: Single Ascending Dose; Part B: Single and Multiple Ascending Dose
Drug: Placebo — Solution for intravenous administration.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of VX-670 at different single and multiple doses in participants with DM1.

ELIGIBILITY:
Key Inclusion Criteria:

- Documented clinical diagnosis of DM1 with age of onset greater than (>) 1 year of age and documented positive genetic test for DM1 in the subject with cytosine thymine guanine (CTG) repeat of at least 100

Key Exclusion Criteria:

- History of any illness or any clinical condition as pre-specified in the protocol

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Parts A and B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) | Part A: From Baseline up to Day 42; Part B: From Baseline and up to Day 168

SECONDARY OUTCOMES:
Part A: Maximum Observed Concentration (Cmax) of VX-670 and its Active Component in Plasma | From Day 1 up to Day 42
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-670 and its Active Component in Plasma | From Day 1 up to Day 42
Part B: Maximum Observed Concentration (Cmax) of VX-670 and its Active Component in Plasma After Each Dose | From Day 1 up to Day 168
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-670 and its Active Component in Plasma After Each Dose | From Day 1 up to Day 168
Part B: Concentration of VX-670 and its Active Component in Muscle | Baseline and at Day 15
Part B: Change in Splicing Index in Muscle Biopsy | Baseline and at Day 15

CONTACTS AND LOCATIONS:
Locations (26):
- United States (8):
  - Stanford Neuromuscular Research, San Carlos, California
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of Kansas Medical Center, Fairway, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University (Sanger Hall), Richmond, Virginia
- Australia (2):
  - Wesley Research Institute, Auchenflower
  - Neuroscience Clinical Trials Unit, Alfred Brain, Melbourne
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven, Belgium
- Canada (5):
  - Hopital de Chicoutimi, Chicoutimi
  - Altasciences Montreal, Montreal
  - McGIll University, Montreal
  - University of Ottawa, Ottawa
  - CHU Research Centre of Quebec, Québec
- Neuromuscular Reference Center Institute of Myology, Paris, France
- Ludwig Maximilians Universitaet Muenchen, München, Germany
- Centro Clinico NeMO, Milan, Italy
- Maastricht University Medical Center, Maastricht, Netherlands
- Hospital Universitario y Politécnico La Fe, Valencia, Spain
- United Kingdom (5):
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - Leonard Wolfson Experimental Neurology Centre CRF, London
  - St. George's University Hospital, London
  - Salford Royal Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/